CLINICAL TRIAL: NCT06766565
Title: QYJD Compound Preparation Promotes Rapid Postoperative Recovery in Early-stage NSCLC Patients by Regulating Tissue Microecology: a Prospective, Randomized Controlled, Open-label, Phase I Clinical Study With Predefined Future Exploration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-026
Record Dates: First submitted 2024-11-15; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: NSCLC
Keywords: QYJD Compound Preparation; clinical trials; rapid rehabilitation; lung tissue microecology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blank control group (No Intervention): Group1 There was no oral drug treatment before surgery. Patients were treated with anti-inflammatory and analgesic therapy postoperatively on a case-by-case basis.
- QYJD Compound Preparation intervention group (Experimental): Group2 In the treatment group, the patients were orally treated with expelling blood stasis and detoxifying compound preparation for 4 days before thoracoscopic radical lung cancer surgery, 2 capsules (0.3g/capsule) at a time, 3 times a day, with lukewarm water, for a total of 4 days.Patients were treated with anti-inflammatory and analgesic therapy postoperatively on a case-by-case basis.
  Interventions: Drug: QYJD Compound Preparation

INTERVENTIONS:
Drug: QYJD Compound Preparation — The intervention group was treated with 2 capsules (g) of expelling stasis and QYJD compound preparation orally for 4 days before thoracoscopic radical surgery for lung cancer, 3 times a day. The blank control group had no oral drug treatment before surgery.
  Arms: QYJD Compound Preparation intervention group

SUMMARY:
QYJD compound preparation has the efficacy of clearing heat and removing toxins, dispelling blood stasis and relieving pain, etc. investigators aimed to explore the effect of expelling blood stasis and removing toxins compound preparation on the microecological changes of lungs of patients with early stage non-small cell lung cancer (NSCLC) by using metagenomics next-generation sequencing (mNGS) technology to carry out a prospective phase I clinical study. The aim of the study was to investigate the effect of the expelling stasis and detoxifying compound preparation on the microecology of lungs of patients with early-stage non-small cell lung cancer (NSCLC), and to conduct a prospective phase I clinical study to provide new ideas for promoting the postoperative rehabilitation of early-stage NSCLC.

DETAILED DESCRIPTION:
1. participants screened for eligibility should sign the appropriate Informed Consent Form (ICF) prior to completing any study procedures.
2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria.

ELIGIBILITY:
Study Population Patients diagnosed with early-stage non-small cell lung cancer in accordance with the Primary Lung Cancer Diagnosis and Treatment Guidelines (2022 Edition) issued by the National Health and Health Commission and the TNM staging criteria of the 8th edition of the International Association for the Study of Lung Cancer (IASLC).

Inclusion criteria:

1. Patients with (a) no contraindications to surgery, early stage NSCLC diagnosed by postoperative pathology, and clinical stage I-IIIA; (b) aged 18-80 years old, with KPS score ≥60; (c) with expected survival of more than 3 months; (d) with no history of smoking; (e) with no previous underlying lung diseases such as bronchiectasis, bronchial asthma, or COPD; (f) without neoadjuvant chemotherapy; (g) with no previous treatment with neoadjuvant chemotherapy; (h) with no previous treatment with neoadjuvant chemotherapy; (i) with no previous treatment with bronchodilatation, bronchial asthma, or COPD; (j) with no previous treatment with neoadjuvant chemotherapy. (f) No neoadjuvant chemotherapy; (g) No history of other systemic malignancies; (h) Sufficient fresh tumor tissue specimens are available.
2. Participants are willing to participate in this study and comply with the study plan;
3. Participants or legally authorized representatives were able to provide written informed consent approved by the ethical review board managing the site.

Exclusion Criteria:

1. the presence of malignant tumors or metastatic foci in other parts of the body;
2. the combination of other organic diseases;
3. psychiatric disorders or communication disorders;
4. lung infections, systemic hematologic diseases, immune system diseases;
5. bronchodilatation, bronchial asthma, or chronic obstructive pulmonary disease and other underlying lung diseases;
6. within the past month, there are antibiotics, immunosuppressive drugs, hormones, probiotics, as well as any those who have taken antibiotics, immunosuppressants, hormones, probiotics, and any form of traditional Chinese medicine or proprietary Chinese medicine within the past month;
7. Those who have a history of smoking;
8. Those who have a history of occupational or environmental exposure to dust, mines, or asbestos.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Rapid rehabilitation indexes | 15 days
  the number of days of postoperative chest drain retention
Rapid rehabilitation indexes | 1 week
  postoperative pain VAS scores
Rapid rehabilitation indexes | 7 day
  six-minute walking experiments
Laboratory indicators of inflammation | through study completion, an average of 1 year
  including white blood cell count, neutrophil count, lymphocyte count, platelet count, NLR, PLR

CONTACTS AND LOCATIONS:
Locations (1):
- Zongyang Yu, Fujian, Fuzhou, China